CLINICAL TRIAL: NCT06817343
Title: An Open-label, Long-term Follow-Up Study to Evaluate the Safety and Tolerability of Gene Therapy With EXG102-031 in Participants With Neovascular Age-related Macular Degeneration
Brief Title: A Long-term Follow up Study of EXG102-031 in Patients With wAMD (Everest LTFU)
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Exegenesis Bio (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EXG102-031-211-LTFU
Record Dates: First submitted 2025-01-30; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Neovascular Age-Related Macular Degeneration (nAMD); Neovascular (Wet) Age-related Macular Degeneration (AMD)
Keywords: EXG102-031; wAMD
MeSH Terms: conditions — Macular Degeneration | interventions — aflibercept

STUDY DESIGN:
Intervention Model Description: Participants from the main study, EXG102-031 (211), will rollover to this study and will be offered Aflibercept IVT PRN to control wAMD symptoms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- All participants who completed the main study of EXG102-031 (Other): All subjects who enroll in this LTFU study have received the experimental treatment with EXG102-031 in the main study, however NO experimental therapy is being administered in this study. The intervention with Aflibercept IVT PRN in this study is NOT experimental.
  Interventions: Biological: Aflibercept (2.0 mg)

INTERVENTIONS:
Biological: Aflibercept (2.0 mg) — PRN IVT Aflibercept

SUMMARY:
In neovascular (wet) age-related macular degeneration (nAMD), the macula, or the part of the eye that provides the clear, detailed central vision, is being affected by abnormal blood vessel growth and leakage. This leakage affects the vision over time and can lead to severe blurriness or blinding. EXG102-031 was made to block the extra vessel formation which would lead to less leakage affecting the vision. Before EXG102-031 can be tested for its efficacy (if it makes vision better), it must be tested to see if it is safely tolerated to confirm it can continue to be studied in more patients with nAMD. This study is designed to fulfill the long-term safety monitoring of EXG102-031. Participants that enroll in this long-term follow-up study have been treated with EXG102-031 under the main study (EXG102-031-211).

DETAILED DESCRIPTION:
Age-related macular degeneration (AMD) is a major cause of blindness and visual impairment in older adults. The wet form of AMD, also called neovascular AMD (nAMD) usually causes faster vision loss than the dry form. The most common current treatments of nAMD are products that inhibit vascular endothelial growth factor (VEGF) (including ranibizumab (LUCENTIS®, Genentech) and aflibercept (EYLEA®, Regeneron) and are delivered by intravitreal injections at 4 to 16 week intervals and continued indefinitely. The Phase I, open-label, multiple-cohort, dose-escalation study designed to evaluate the safety and tolerability of EXG102-031 gene therapy in subjects with previously treated nAMD (EXG102-031-211). In the main study safety was assessed over 52 weeks after the administration of EXG102-031. This long-term follow-up study will assess safety for an additional 36 months for all participants enrolled in the main study. Participants will return to the clinic regularly for ocular assessments including assessment of whether supplemental therapy with aflibercept is needed.

ELIGIBILITY:
Inclusion Criteria:

* Must have been previously enrolled in the parent study (EXG102-031-211) and must have received subretinal EXG102-031 in the parent study;
* Are willing and able to sign the study written informed consent form;
* Must be willing and able to comply with all study procedures.

There are no exclusion Criteria in this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Evaluation of long-term safety by measuring frequency, type, and intensity of ocular and non-ocular adverse events (AEs) and serious adverse events (SAEs) through Month 36 (Year 4) post EXG102-031 administration. | Month 36

SECONDARY OUTCOMES:
Evaluation of potential efficacy by measuring change from baseline in best corrected visual acuity (BCVA) measured using the ETDRS method and average number of doses of aflibercept supplemental therapy through Month 36 (Year 4) | Month 36

OTHER OUTCOMES:
Anatomical characteristics of EXG102-031 by measuring the change from baseline in central retinal thickness as measured by SD-OCT at Month 36 (Year 4) | Month 36
Pharmacodynamic characteristics of EXG102-031 by measuring the transgene expression in aqueous fluid at Month 36 (Year 4) | Month 36

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Sierra Eye Associates, Reno, Nevada
  - Erie Retina Research, Erie, Pennsylvania

IPD SHARING:
Plan to Share IPD: No